CLINICAL TRIAL: NCT02214199
Title: Effectiveness of Cervicothoracic Manipulative Treatment in Unilateral Shoulder Impingement Syndrome: A Randomized Controlled Trial.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Collaborators: Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD (Lecturer), Universidad de Almeria
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 21/2013
Record Dates: First submitted 2014-08-09; First posted 2014-08-12 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Shoulder Pain; Manual Theapy; Exercises Therapy
Keywords: Shoulder Pain; Shoulder Impingement Syndrome; Exercise therapy; Randomized Controlled Trial
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Therapy (Active Comparator): Home exercises for 30 minutes (2/weeks) with muscle stretching and strengthening the shoulder girdle.
  Interventions: Other: Home Exercises
- Manipulative Therapy Techniques (Experimental): Lift Technique for mid-thoracic spine. Mobilization by low cervical spine on the upper lateral thoracic translation. Technical Dog flexion for high thoracic spine (T1-T4). Technical Dog flexion for mid-thoracic spine (T5-T8). Technical Dog flexed to low thoracic spine (T9-T12). Direct drive technology prone to mid-thoracic spine.
  Interventions: Other: Manipulative Therapy Techniques

INTERVENTIONS:
Other: Manipulative Therapy Techniques
  Arms: Manipulative Therapy Techniques
Other: Home Exercises
  Arms: Exercise Therapy

SUMMARY:
The objective of this protocol is to compare degree of improvement can be achieved in patients with shoulder pain by treatment with Manipulative Techniques for the cervicothoracic spine versus home exercises.

DETAILED DESCRIPTION:
Design: Randomized Clinical Trial. Objective: to determine the effects of manipulative techniques for the ervicothoracic spine versus home exercises on pain, disability, and range of movement in patients with unilateral shoulder inmingement syndrome.

Methods and Measures: ninety-two subjects will be randomly assigned to one of two groups.

Intervention: For 5-weeks, the groups 1 will undergo tratment comprising manipulative protocol techniques for the cervicothoracic spine (2/week) and the group 2 will develop a home exercise (2/week).

Main Outcome Measures: Intensity of pain, disability, and range of motion data will be collected at baseline, and 24hr after the last therapy application. Mixed-model analyses of variance will be used to examine the effects of the treatment on each outcome measure.

ELIGIBILITY:
Inclusion Criteria:

1. Report of pain or dysfunction with overhead activities
2. Demonstration of pain during active shoulder movements
3. Demonstration of a positive Neer/Hawkins-Kennedy test
4. Recent onset within the last 12 months
5. Report of non-traumatic onset
6. Demonstration of a painful arc of the arm from 60° to 120° of flexion
7. Report of a baseline pain level of ≥2/10 on an 11 point numeric scale

Exclusion Criteria:

* The presence of any red flags
* A history of frozen shoulder
* Disorders of the acromioclavicular joint
* Degenerative arthritis of the glenohumeral joint
* Known calcifying tendonitis (if identified by radiograph)
* Shoulder instability
* Posttraumatic disorders
* Shoulder surgery and/or elbow, hand, wrist and blatantly misdiagnosed cervical spine disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Disability Questionnaire Arm, Shoulder and Hand (DASHe) | At baseline and 5 weeks
  This questionnaire asks about the symptoms as well as your ability to perform certain activities. This questionnaire has 30 items, and the results are clasified in: no difficulty, mild difficulty, moderate dificulty, severe dificulty and unable

SECONDARY OUTCOMES:
Shoulder Disability Questionnaire | At baseline and 5 weeks
  Shoulder Disability Questionnaire is a mesure covering 16 items designed to evaluate functional status limitation in patients with shoulder disorders.
Hawkins-Kennedy Test | At baseline and 5 weeks
  The Hawkins and Kennedy test was interpreted as indicative of impingement between the greater tuberosity of the humerus against the coraco- humeral ligament, trapping all those structures which intervene. It has been reported as less reliable than the Neer impingement test.
Neer Test. | At baseline and 5 weeks
  Neer's Test assesses for possible rotator cuff impingement. Stabilize the scapula and with the thumb pointing down and passively flex the arm. Pain is a positive test.
Range of Motion | At baseline and 5 weeks
  The range of motion will be evaluated in flexion, extension, rotation, adduction, and abduction.
Visual Analogue Scale | At baseline and 5 weeks
  A 10-point numerical pain scale (0:no pain, 10: maximum pain) assesses the intensity of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Almeria, Almería, Almería, Spain

REFERENCES:
- [Background] Rhon DI, Boyles RB, Cleland JA. One-year outcome of subacromial corticosteroid injection compared with manual physical therapy for the management of the unilateral shoulder impingement syndrome: a pragmatic randomized trial. Ann Intern Med. 2014 Aug 5;161(3):161-9. doi: 10.7326/M13-2199. PMID 25089860
- [Background] Cook C, Learman K, Houghton S, Showalter C, O'Halloran B. The addition of cervical unilateral posterior-anterior mobilisation in the treatment of patients with shoulder impingement syndrome: a randomised clinical trial. Man Ther. 2014 Feb;19(1):18-24. doi: 10.1016/j.math.2013.05.007. Epub 2013 Jun 20. PMID 23791561
- [Background] Alburquerque-Sendin F, Camargo PR, Vieira A, Salvini TF. Bilateral myofascial trigger points and pressure pain thresholds in the shoulder muscles in patients with unilateral shoulder impingement syndrome: a blinded, controlled study. Clin J Pain. 2013 Jun;29(6):478-86. doi: 10.1097/AJP.0b013e3182652d65. PMID 23328323
- [Background] Maenhout AG, Mahieu NN, De Muynck M, De Wilde LF, Cools AM. Does adding heavy load eccentric training to rehabilitation of patients with unilateral subacromial impingement result in better outcome? A randomized, clinical trial. Knee Surg Sports Traumatol Arthrosc. 2013 May;21(5):1158-67. doi: 10.1007/s00167-012-2012-8. Epub 2012 May 12. PMID 22581193
- [Background] Camargo PR, Avila MA, Alburquerque-Sendin F, Asso NA, Hashimoto LH, Salvini TF. Eccentric training for shoulder abductors improves pain, function and isokinetic performance in subjects with shoulder impingement syndrome: a case series. Rev Bras Fisioter. 2012 Jan-Feb;16(1):74-83. doi: 10.1590/s1413-35552012000100013. PMID 22441232
- [Background] Hidalgo-Lozano A, Fernandez-de-las-Penas C, Diaz-Rodriguez L, Gonzalez-Iglesias J, Palacios-Cena D, Arroyo-Morales M. Changes in pain and pressure pain sensitivity after manual treatment of active trigger points in patients with unilateral shoulder impingement: a case series. J Bodyw Mov Ther. 2011 Oct;15(4):399-404. doi: 10.1016/j.jbmt.2010.12.003. Epub 2011 Jan 17. PMID 21943613
- [Background] Gwilym SE, Oag HC, Tracey I, Carr AJ. Evidence that central sensitisation is present in patients with shoulder impingement syndrome and influences the outcome after surgery. J Bone Joint Surg Br. 2011 Apr;93(4):498-502. doi: 10.1302/0301-620X.93B4.25054. PMID 21464489
- [Background] Koike Y, Sano H, Kinjyo T, Imamura I, Masahiro O, Goto M, Ooyama M, Kita A, Itoi E. Shoulder surface temperature and bone scintigraphy findings in patients with rotator cuff tears. Ups J Med Sci. 2011 May;116(2):142-7. doi: 10.3109/03009734.2010.545150. Epub 2011 Feb 16. PMID 21323485
- [Background] Hidalgo-Lozano A, Fernandez-de-las-Penas C, Alonso-Blanco C, Ge HY, Arendt-Nielsen L, Arroyo-Morales M. Muscle trigger points and pressure pain hyperalgesia in the shoulder muscles in patients with unilateral shoulder impingement: a blinded, controlled study. Exp Brain Res. 2010 May;202(4):915-25. doi: 10.1007/s00221-010-2196-4. Epub 2010 Feb 26. PMID 20186400
- [Background] Osteras H, Torstensen TA. The dose-response effect of medical exercise therapy on impairment in patients with unilateral longstanding subacromial pain. Open Orthop J. 2010 Jan 5;4:1-6. doi: 10.2174/1874325001004010001. PMID 20148093